CLINICAL TRIAL: NCT03555188
Title: A Randomised, Placebo Controlled Trial to Determine the Efficacy and Mode of Action of Ondansetron in the Treatment of Irritable Bowel Syndrome With Diarrhoea
Brief Title: TReatment of Irritable Bowel Syndrome With Diarrhoea Using Titrated ONdansetron Trial
Acronym: TRITON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: Barnsley Hospital NHS Foundation Trust (Other); Barts & The London NHS Trust (Other); County Durham and Darlington NHS Foundation Trust (Other Government); Flinders University (Other); The Leeds Teaching Hospitals NHS Trust (Other); London North West Healthcare NHS Trust (Other); NHS Lothian (Other Government); Queen Mary University of London (Other); Sandwell & West Birmingham Hospitals NHS Trust (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other); University College London Hospitals (Other); University Hospitals of North Midlands NHS Trust (Other); Manchester University NHS Foundation Trust (Other Government); University of Manchester (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15/74/01
Record Dates: First submitted 2018-04-18; First posted 2018-06-13 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: IBS - Irritable Bowel Syndrome
Keywords: Diarrhoea
MeSH Terms: conditions — Irritable Bowel Syndrome; Diarrhea | interventions — Ondansetron

STUDY DESIGN:
Intervention Model Description: TRITON is a parallel group, randomised, double-blinded, placebo controlled trial, to determine the superiority of Ondansetron.
Who Masked: Participant, Investigator
Masking Description: This is a double-blinded study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ondansetron (Experimental): Taken orally 4mg-24mg daily for 12 weeks. Dose to be amended throughout according to symptoms.
  Interventions: Drug: Ondansetron
- Placebo (Placebo Comparator): Taken orally 4mg-24mg daily for 12 weeks. Dose to be amended throughout according to symptoms.
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Drug: Ondansetron — Ondansetron is a highly selective receptor antagonist (5-HT3RA)

SUMMARY:
A placebo controlled study to determine the efficacy and mode of action of ondansetron in the treatment of irritable bowel syndrome with diarrhoea.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) affects around 10% of the population and accounts for 1.8 million consultations/year in primary care in England and Wales (0.6 million patients). Around one third of patients meet the criteria for IBS with diarrhoea (IBS-D) and despite its high prevalence, there is no satisfactory treatment at present. Loperamide is currently used to reduce bowel frequency, however it does not improve symptoms such abdominal pain.

Other symptoms of IBS-D include frequent, loose, or watery stools with associated urgency, which can severely limit socialising, travelling, and eating out, resulting in a reduced quality of life and work productivity.

The primary aim of the study is to determine the effectiveness and safety of the use of ondansetron in patients with the symptoms of IBS-D including urgency, looseness of stool, frequency of defecation and abdominal discomfort. Ondansetron belongs to a class of drug known as 5HT3RAs and a recent meta-analysis shows that 5HT3RAs is an effective treatment for IBS-D, improving stool consistency and reducing frequency and urgency of defecation.

400 patients with IBS-D will be randomised on a 1:1 basis to receive either Ondansetron or Placebo. Both treatments will be administered in oral doses of between 4-24mg daily for 12 weeks. Dose titration will be undertaken in the first two weeks of the study to avoid constipation.

The primary outcome of response will be assessed at 12 weeks post randomisation using patient reported data on daily stool frequency and abdominal pain.

If ondansetron is effective in the trial, it could easily be widely adopted since it is an inexpensive, safe, and generic drug. By providing an effective treatment, it could not only reduce patient symptoms, but also reduce costs of repeated referral and investigation.

ELIGIBILITY:
Inclusion Criteria:

1. Written (signed and dated) informed consent.
2. Considered fit for study participation.
3. Meeting Rome IV criteria for IBS-D
4. Aged ≥ 18 years
5. Undergone standardised workup to exclude the following alternative diagnoses:

   1. Microscopic colitis (colonoscopy or flexible sigmoidoscopy),
   2. Bile acid diarrhoea (SeHCAT results of > 10%, C4 results of <19 ng/ml or failed 1 week trial of a bile acid binding agent [colestyramine 4g t.d.s. , colesevelam 625mg t.d.s. or equivalent]) within previous 5 years, Note: Cholecystectomy will not be an exclusion criteria if bile acid diarrhoea has been excluded. Patients with SeHCAT values of 5-10% will be eligible if they fail to respond to a 1 week trial of bile acid binding agent (see above)
   3. Lactose malabsorption.
   4. Coeliac disease (tTG or duodenal biopsy)
6. Patients of child bearing potential or with partners of child bearing potential must agree to use methods of medically acceptable forms of contraception during the study and for 90 days after completion of study drug, (e.g. implants, injectable, combined oral contraceptives, barrier methods, true abstinence (when this is in line with the preferred and usual lifestyle of the patient) or vasectomised partners).
7. For women of child bearing potential, a negative pregnancy test should be performed within 72 hours of confirmation of eligibility.
8. Weekly average worst pain score >= X on a 0 to 100 point scale <<redacted to prevent patient bias>>.
9. Any stools with a consistency of X on the Bristol Stool Form score (BSFS) for X day per week<<redacted to prevent patient bias>>.

Exclusion Criteria:

1. Gastrectomy
2. Intestinal resection
3. Other known organic GI diseases (e.g. Inflammatory bowel disease - Crohns disease, Ulcerative colitis.)
4. Unable or unwilling to stop restricted medication including regular loperamide, antispasmodics (e.g. buscopan, mebeverine, peppermint oil, alverine citrate), eluxadoline, tricyclic antidepressant doses >30mg/day or other drugs likely in the opinion of the investigator to alter bowel habit. These medicines should be discontinued for a 7 day washout period prior to registration. Note: Intermittent loperamide will be permitted but only as rescue medication
5. QTc interval ≥450msec for men and ≥470msec for women. Assessed within the last 3 months by a 12-lead ECG.
6. Previous chronic use of ondansetron or contraindications to it (rare as per BNF)
7. Pulse, Blood pressure, FBC or LFTs outside the normal ranges according to the site's local definition of normal. Assessed within the last 3 months.Note: Minor rises in ALT (<2 x upper limit of normal) will be acceptable but the patient's GP will be informed if they remain elevated at end of the study.
8. Women who are pregnant or breastfeeding
9. Patients currently participating or who have been in an IMP trial in the previous three months where the use of the IMP may cause issues with the assessment of causality in this study.
10. Currently taking SSRIs or tricyclic antidepressants (unless at a stable dose for at least 3 months and with no plan to change the dose during the study).
11. Currently taking and unwilling or unable to stop any of the prohibited medications.*

    *Prohibited medications - Apomorphine & tramadol which interact with ondansetron. Caution should be taken with patients on QT prolonging drugs and cardio toxic drugs. These patients should be reviewed by the PI to determine if they are suitable for the study.
12. Patients with stools of consistency X on the Bristol Stool Form score (BSFS) for X days a week <<redacted to prevent patient bias>>.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Weekly responder for abdominal pain and stool consistency | 12 weeks
  Measured at 12 weeks post randomisation and defined, as recommended by the FDA, as patient being a weekly responder for BOTH pain intensity AND stool consistency for at least 6 weeks in the 12 week treatment period.

SECONDARY OUTCOMES:
Stool Frequency | 12 weeks
  For the endpoint analysis, the mean number of stools per day over the last month (weeks 9-12) will be used.
Stool Consistency | 12 weeks
  Defined as number of days per week with at least 1 loose stool and the average stool consistency over the last month (weeks 9-12)
Urgency of defecation | 12 weeks
  The mean daily urgency score over last month (weeks 9-12)
Satisfactory relief of IBS symptoms | 12 weeks c
  Defined as satisfactory relief of IBS symptoms for at least 6 out of 12 weeks
Functional dyspepsia | This information is collected via a questionnaire which asks the patient about any symptoms associated with IBS that they may be experiencing. This information is collected at baseline (week 0) and again after treatment (week 12).
  SF-LDQ questionnaire at week 0 and week 12
IBS Symptom Severity Scale | This information is collected at baseline (week 0) and again after treatment (week 12).
  Irritable Bowel Syndrome Symptom Severity Scale questionnaire which asks patients about their IBS symptoms such as abdominal pain etc. The patients will provide yes/no answer or a score on a 0-100 scale with 0 being the minimum amount and 100 being define as quite severe/definitely.
Rescue Medication | 12 weeks
  The total number of days taken loperamide throughout the 12 weeks
Abdominal pain score | 12 weeks
  The mean daily pain score over the last month (weeks 9-12)
Hospital Anxiety and Depression Scale | This information is collected at baseline (week 0) and again after treatment (week 12).
  Hospital Anxiety and Depression Scale questionnaire. This information is collected via a questionnaire which asks the patient about their general overall feelings. It asks a variety of question and the patient is to tick the box beside the reply that is closest to how they feel. Each question has 1 of 4 potential replies (feelings) that vary depending on the nature of the question.
IBS Quality of life summary score | This information is collected via a questionnaire which asks the patient about the quality of their life. This information is collected at baseline (week 0) and again after treatment (week 12).
  IBS-QOL questionnaire at 0 and 12 weeks
Stool frequency post treatment | 4 weeks
  The mean number of stools per day for 1 months after treatment (weeks 13-16)
Stool consistency post treatment | 4 weeks
  The mean daily stool consistency over 1 month (weeks 13-16) .
Urgency of defecation post treatment | 4 weeks
  The mean daily urgency score over 1 month post treatment (weeks 13-16).
Abdominal pain post treatment | 4 weeks
  The mean daily pain score over 1 month (weeks 13-16)

OTHER OUTCOMES:
Colonic transit | 12 weeks
  Colonic Transit study to determine if ondansetron slows colonic transit.
Ondansetron and cyclical retrograde propagated contractions in the sigmoid colon | 12 weeks
  High resolution colonic manometry at baseline and week 12
Ondansetron and rectal compliance/pressure thresholds for pain/urgency. | 12 weeks
  Barostat assessment at baseline and week 12
Does ondansetron reduce total faecal bile acids and total tryptase and does the reduction correlate with changes in urgency? | 12 weeks
  Stool samples collected at baseline and week 12
Do polymorphisms in the TPH-1 gene predict response to ondansetron and does this alter 5-HT or TPH1-mRNA | 12 weeks
  Bloods and biopsies taken at baseline and week 12

CONTACTS AND LOCATIONS:
Overall Officials: Robin Spiller, Study Chair — University of Nottingham
Locations (14):
- United Kingdom (14):
  - Barnsley Hospital NHS Foundation Trust, Barnsley
  - Sandwell and West Birmingham Hospitals NHS Trust, Birmingham
  - County Durham and Darlington NHS Foundation Trust, Durham
  - Westen General Hosptal, Edinburgh, Edinburgh
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - London North West NHS Foundation Trust, London
  - Queen Mary, University of London, London
  - University College London Hospitals NHS Foundation Trust, London
  - Salford Royal Hospital, Manchester
  - University Hospital of South Manchester, Manchester
  - SouthTees Hospitals NHS FoundationTrust, Middlesbrough
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Royal Hallamshire Hospital, Sheffield
  - University Hospitals of North Midlands NHS Trust, Stoke

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gunn D, Topan R, Barnard L, Fried R, Holloway I, Brindle R, Corsetti M, Scott M, Farmer A, Kapur K, Sanders D, Eugenicos M, Trudgill N, Whorwell P, Mclaughlin J, Akbar A, Houghton L, Dinning PG, Aziz Q, Ford AC, Farrin AJ, Spiller R. Randomised, placebo-controlled trial and meta-analysis show benefit of ondansetron for irritable bowel syndrome with diarrhoea: The TRITON trial. Aliment Pharmacol Ther. 2023 Jun;57(11):1258-1271. doi: 10.1111/apt.17426. Epub 2023 Mar 3. PMID 36866724